CLINICAL TRIAL: NCT02578524
Title: Satisfaction With Multifocal vs Accommodating Lens Implants 2 Years After Surgery
Status: Completed | Type: Observational
Sponsor: MDbackline, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: BAU141212
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Cataract
Keywords: cataract satisfaction
MeSH Terms: conditions — Cataract | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Accommodating Lenses: Patients who underwent surgery with an accommodating lens implant.
  Interventions: Other: Survey
- Multifocal Lenses: Patients who underwent surgery with an multifocal lens implant.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
This study will examine patient satisfaction and spectacle independence using a survey in patients who have undergone uncomplicated cataract surgery with a presbyopia-correcting lens at least 2 years prior to administration of the survey.

DETAILED DESCRIPTION:
Purpose: To compare patient-reported satisfaction with a multifocal vs an accommodating presbyopia-correcting at least two years following implantation of either type of implant.

Number of study subjects: 200 (half with multifocal and half with accommodating lens implants)

In this study, we will send a secure, online questionnaire to patients who have previously undergone cataract surgery at least two years previously. Patients will receive an email invitation, and by clicking the embedded link and verifying their identity with date of birth and phone number, they will be directed to a survey. The survey will ask the following types of questions:

* overall satisfaction with the surgery
* would they do the same surgery again?
* would they choose the same (elective) lens implant again?
* for what types of activities (reading newspaper, driving, driving at night, fine print) do they require glasses to see clearly?
* do they experience glare and halo symptoms?
* how bothered is the patient by these symptoms?

These data will be stored on a secure server. Statistical analysis will be done by a statistician, using a student's t-test to determine statistical significance of any difference between patients with different types of lens implants.

No intervention will be planned with patients, other than analyzing the survey results. All patient identifying (demographic) information will be carefully protected according to HIPAA and HITECH standards.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncomplicated bilateral cataract surgery with either multifocal or accommodating lens implants performed at least 24 months previously
* Patients with or without astigmatic keratotomy or other simultaneous procedures may be included, so long as exclusion criteria are not met.

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that, in the best judgment of the investigator, could affect their satisfaction with surgery
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.)
* Patients with ≥ grade 1 posterior capsule opacity at their last visit

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent cataract surgery with a multifocal or accommodating lens implant at least two years prior to the survey.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Satisfaction | At least 24 months after cataract surgery was performed. No upper limit on time since surgery.
  The patients will be asked to rate their satisfaction with their surgical results on a scale of "very satisfied", "satisfied", "neither satisfied nor dissatisfied", "dissatisfied", or "very dissatisfied".

SECONDARY OUTCOMES:
Ability to drive without glasses | At least 24 months after cataract surgery was performed. No upper limit on time since surgery.
  The patients will be asked to rate their ability to drive without glasses on a scale of "very satisfied", "satisfied", "neither satisfied nor dissatisfied", "dissatisfied", or "very dissatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — MDbackline, LLC
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States